CLINICAL TRIAL: NCT00710333
Title: A Single-centre, Double Blind, Randomised, Tolerance Study to Investigate the Safety of Juvista 500ng/100µL/Linear cm When Administered Following Excision of Ear Lobe Keloids.
Brief Title: Safety of Juvista When Administered Following Excision of Ear Lobe Keloids
Acronym: RN1001-0093
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Amanda Hilton Senior Clinical Research Manager, Renovo Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1001-0093
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): 500ng dose
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: Avotermin

INTERVENTIONS:
Drug: Avotermin — 10 patients undergoing surgical revision of bilateral keloids will be dosed with 500ng Juvista/100µL per cm of wound margin to one ear lobe and placebo to the other and followed up for three months after dosing to assess the local and systemic tolerability.
  Arms: 2
Drug: placebo — placebo
  Arms: 1

SUMMARY:
This trial will assess the safety and efficacy of 500ng Juvista per linear cm of wound margin administered by intradermal injection following the excision of keloid scars on the ear lobe. Ear lobe keloids commonly occur after ear piercing and can be particularly distressing for patients as they are very difficult to conceal and are usually bilateral. As the recurrence rate and growth rate of keloids can vary significantly between individuals, trial subjects will have bilateral ear lobe keloids and will act as their own control. One ear lobe will be treated with Juvista following keloid excision and one with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years who have given written informed consent.
* Patients with bilateral ear lobe keloid scars suitable for surgical excision which will result in a single wound on each ear lobe no greater than 2cm long and restricted to the skin, fat and fibrous tissue of the ear lobe.
* Patients with, in the opinion of the investigator, clinically acceptable results for the laboratory tests specified in the trial protocol (see Protocol Section 6.3.2). All laboratory tests must be performed within 28 days of the first trial dose administration.
* Female patients of child bearing potential who are using a highly effective method(s) of contraception and agree to do so from at least the screening visit until one month after administration of the final study dose. For the purposes of the protocol, highly effective method(s) of contraception will be defined as consistently and correctly used implants, injectables, combined oral contraceptives, sexual abstinence or a vasectomised partner.

Exclusion Criteria:

* Patients who have had ear lobe keloids treated with irradiation, cryosurgery, corticosteriods, or other pharmacological agents in the three months prior to the first trial dose administration.
* Patients with a history of a bleeding disorder.
* Patients who on direct questioning and/or physical examination have past or present evidence of eczema or psoriasis local to the site of administration, uncontrolled diabetes (fasting plasma glucose concentration consistently at or above 7.0mmol 1-1 (126 mg dl-1), severely immunocompromised patients and/or malignant skin tumours e.g. melanomas, squamous or basal cell carcinomas.
* Patients with a skin disorder, not related to the keloid disease, that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Patients with a history of malignancy in the last 5 years.
* Patients with a history of hypersensitivity to any of the drugs or dressings used in this trial.
* Patients who are taking, or have taken any investigational product or participated in a clinical trial in the three months prior to first trial dose administration.
* Patients undergoing investigations or changes in management for an existing medical condition.
* Patients who, in the opinion of the Investigator, are unlikely to complete the trial for whatever reason.
* Female patients who are pregnant or lactating.
* Patients with a creatinine clearance (CLcr) of 80ml/min or less. Creatinine clearance will be determined from the serum creatinine level at pre-study screening using the following formula.
* CLcr = (140-age (years)) x weight (kg)/ 72 x serum creatinine (mg/dL) { x 0.85 for females}
* Patients who are not able to undergo MRI scanning due to their medical history or Physical condition.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse events | 3 months

SECONDARY OUTCOMES:
Keliod recurrence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: V V Young, MD, Principal Investigator — Body Aesthetic Plastic Surgery and Skincare Center
Locations (1):
- Body Aesthetic Plastic Surgery and Skincare Center, St Louis, Missouri, United States